CLINICAL TRIAL: NCT02958111
Title: Single-agent Capecitabine as Adjuvant Chemotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma: A Phase 3, Multicentre, Randomised Controlled Trial (CAN)
Brief Title: Single-agent Capecitabine as Adjuvant Chemotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma
Acronym: CAN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Peking University (Other); Air Force Military Medical University, China (Other); Second Affiliated Hospital of Soochow University (Other); West China Hospital (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other); First People's Hospital of Foshan (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Cancer Hospital of Guizhou Province (Other); Xiangya Hospital of Central South University (Other); First Affiliated Hospital of Zhejiang University (Other); Jilin Provincial Tumor Hospital (Other); Henan Cancer Hospital (Other Government); Hunan Cancer Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Prof, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-FXY-075
Record Dates: First submitted 2016-10-26; First posted 2016-11-08 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Adjuvant chemotherapy; Capecitabine
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant capecitabine (Experimental): Adjuvant chemotherapy with single-agent capecitabine
  Interventions: Drug: Capecitabine
- Observation (No Intervention): Clinical follow-up and surveillance only

INTERVENTIONS:
Drug: Capecitabine — Patients will receive capecitabine (650 mg/m2 bid, p.o.，d1-21，q3wks; continued until disease progression, unacceptable toxicity, or over 1 year).
  Arms: Adjuvant capecitabine

SUMMARY:
This is an randomized, controlled, multicenter phase 3 clinical trial. The purpose of this study is to evaluate the efficacy and safety of single-agent capecitabine as adjuvant chemotherapy in locoregionally advanced nasopharyngeal carcinoma (NPC).

DETAILED DESCRIPTION:
In this study, NPC patients (stage III-IV A, except T3-4 N0 and T3 N1) who finished the curative radiotherapy will be randomized to the observation group and capecitabine group (650 mg/m2 bid, p.o.，d1-21，q3wks; continued until disease progression, unacceptable toxicity, or over 1 year). The primary endpoint is progression-free survival (PFS). Secondary end points include overall survival (OS), distant failure-free survival (D-FFS), locoregional failure-free survival (LR-FFS), toxic effects, and quality of life (QOL). All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Performance status of Eastern Cooperative Oncology Group (ECOG) grade 0 or 1
3. Tumor staged as American Joint Committee on Cance (AJCC) III-IV A (except T3-4 N0, T3 N1), with newly histologically confirmed non-keratinizing NPC
4. Within 12-16weeks after completion of the recommended curative radiotherapy treatment
5. No clinical evidence of persistent loco-regional disease or distant metastases after radiotherapy
6. Complete the recommended concurrent chemotherapy ± induction chemotherapy
7. Adequate hematologic (neutrophil count > 1.5×10^9/L, hemoglobin > 90g/L and platelet count > 100×10^9/L), hepatic (alanine aminotransferase, aspartate aminotransferase ≤ 1.5×ULN, bilirubin ≤ 1.5×ULN, alkaline phosphatase < 2.5×ULN) and renal function (creatinine clearance > 50 ml/min)
8. Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

1. Patients who could not tolerate or allergic to capecitabine.
2. Illness that would interfere with oral medication, including dysphagia, chronic diarrhea, or ileus
3. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
4. Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
5. Patients who received surgery treatment, biotherapy or immunotherapy during or before radiotherapy.
6. Patients who are receiving or highly likely to receive other chemotherapy treatment, biotherapy or immunotherapy.
7. History of previous radiotherapy before the curative radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).
8. Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes before the curative radiotherapy
9. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2017-01; Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years
Distant failure-free survival | 3 years
Locoregional failure-free survival | 3 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year
Quality of life (QOL) as assessed by EORTC quality of life questionnaire(QLQ)-C30 | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu YC, Wang WY, Twu CW, Jiang RS, Liang KL, Wu CT, Lin PJ, Huang JW, Hsieh HY, Lin JC. Prognostic impact of adjuvant chemotherapy in high-risk nasopharyngeal carcinoma patients. Oral Oncol. 2017 Jan;64:15-21. doi: 10.1016/j.oraloncology.2016.11.008. Epub 2016 Nov 30. PMID 28024719
- [Background] Twu CW, Wang WY, Chen CC, Liang KL, Jiang RS, Wu CT, Shih YT, Lin PJ, Liu YC, Lin JC. Metronomic adjuvant chemotherapy improves treatment outcome in nasopharyngeal carcinoma patients with postradiation persistently detectable plasma Epstein-Barr virus deoxyribonucleic acid. Int J Radiat Oncol Biol Phys. 2014 May 1;89(1):21-9. doi: 10.1016/j.ijrobp.2014.01.052. PMID 24725686
- [Background] Blanchard P, Lee A, Marguet S, Leclercq J, Ng WT, Ma J, Chan AT, Huang PY, Benhamou E, Zhu G, Chua DT, Chen Y, Mai HQ, Kwong DL, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Zhang L, Hui EP, Lu TX, Bourhis J, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy and radiotherapy in nasopharyngeal carcinoma: an update of the MAC-NPC meta-analysis. Lancet Oncol. 2015 Jun;16(6):645-55. doi: 10.1016/S1470-2045(15)70126-9. Epub 2015 May 6. PMID 25957714
- [Background] Ribassin-Majed L, Marguet S, Lee AWM, Ng WT, Ma J, Chan ATC, Huang PY, Zhu G, Chua DTT, Chen Y, Mai HQ, Kwong DLW, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Bourhis J, Pignon JP, Blanchard P. What Is the Best Treatment of Locally Advanced Nasopharyngeal Carcinoma? An Individual Patient Data Network Meta-Analysis. J Clin Oncol. 2017 Feb 10;35(5):498-505. doi: 10.1200/JCO.2016.67.4119. Epub 2016 Dec 5. PMID 27918720
- [Background] Stockler MR, Harvey VJ, Francis PA, Byrne MJ, Ackland SP, Fitzharris B, Van Hazel G, Wilcken NR, Grimison PS, Nowak AK, Gainford MC, Fong A, Paksec L, Sourjina T, Zannino D, Gebski V, Simes RJ, Forbes JF, Coates AS. Capecitabine versus classical cyclophosphamide, methotrexate, and fluorouracil as first-line chemotherapy for advanced breast cancer. J Clin Oncol. 2011 Dec 1;29(34):4498-504. doi: 10.1200/JCO.2010.33.9101. Epub 2011 Oct 24. PMID 22025143
- [Background] Simkens LH, van Tinteren H, May A, ten Tije AJ, Creemers GJ, Loosveld OJ, de Jongh FE, Erdkamp FL, Erjavec Z, van der Torren AM, Tol J, Braun HJ, Nieboer P, van der Hoeven JJ, Haasjes JG, Jansen RL, Wals J, Cats A, Derleyn VA, Honkoop AH, Mol L, Punt CJ, Koopman M. Maintenance treatment with capecitabine and bevacizumab in metastatic colorectal cancer (CAIRO3): a phase 3 randomised controlled trial of the Dutch Colorectal Cancer Group. Lancet. 2015 May 9;385(9980):1843-52. doi: 10.1016/S0140-6736(14)62004-3. Epub 2015 Apr 7. PMID 25862517
- [Background] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945
- [Background] Zhang L, Huang Y, Hong S, Yang Y, Yu G, Jia J, Peng P, Wu X, Lin Q, Xi X, Peng J, Xu M, Chen D, Lu X, Wang R, Cao X, Chen X, Lin Z, Xiong J, Lin Q, Xie C, Li Z, Pan J, Li J, Wu S, Lian Y, Yang Q, Zhao C. Gemcitabine plus cisplatin versus fluorouracil plus cisplatin in recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 trial. Lancet. 2016 Oct 15;388(10054):1883-1892. doi: 10.1016/S0140-6736(16)31388-5. Epub 2016 Aug 23. PMID 27567279
- [Background] Hui EP, Ma BB, Leung SF, King AD, Mo F, Kam MK, Yu BK, Chiu SK, Kwan WH, Ho R, Chan I, Ahuja AT, Zee BC, Chan AT. Randomized phase II trial of concurrent cisplatin-radiotherapy with or without neoadjuvant docetaxel and cisplatin in advanced nasopharyngeal carcinoma. J Clin Oncol. 2009 Jan 10;27(2):242-9. doi: 10.1200/JCO.2008.18.1545. Epub 2008 Dec 8. PMID 19064973
- [Derived] Liu Y, Yan W, Chen Y, Miao J, Zhang H, Wang J, Zhang Y, Huang X, Wang K, Qu Y, Chen X, Zhang J, Luo J, Li YX, Zhao C, Ma J, Wu R, Yi J. Treatment response-adapted risk index model for survival prediction and adjuvant chemotherapy selection in nonmetastatic nasopharyngeal carcinoma. NPJ Digit Med. 2025 Sep 1;8(1):564. doi: 10.1038/s41746-025-01918-2. PMID 40890288
- [Derived] He Q, Luo X, Liu L, Zhao C, Li Z, Jin F. Effect of immune-modulating metronomic capecitabine as an adjuvant therapy in locoregionally advanced nasopharyngeal carcinoma. BMC Immunol. 2024 May 6;25(1):28. doi: 10.1186/s12865-024-00621-3. PMID 38710996
- [Derived] Chen YP, Liu X, Zhou Q, Yang KY, Jin F, Zhu XD, Shi M, Hu GQ, Hu WH, Sun Y, Wu HF, Wu H, Lin Q, Wang H, Tian Y, Zhang N, Wang XC, Shen LF, Liu ZZ, Huang J, Luo XL, Li L, Zang J, Mei Q, Zheng BM, Yue D, Xu J, Wu SG, Shi YX, Mao YP, Chen L, Li WF, Zhou GQ, Sun R, Guo R, Zhang Y, Xu C, Lv JW, Guo Y, Feng HX, Tang LL, Xie FY, Sun Y, Ma J. Metronomic capecitabine as adjuvant therapy in locoregionally advanced nasopharyngeal carcinoma: a multicentre, open-label, parallel-group, randomised, controlled, phase 3 trial. Lancet. 2021 Jul 24;398(10297):303-313. doi: 10.1016/S0140-6736(21)01123-5. Epub 2021 Jun 7. PMID 34111416